CLINICAL TRIAL: NCT03599427
Title: Added Value of Systemic Lidocaine in Combination With Local Infiltration Analgesia for Knee Arthroscopic Procedures
Brief Title: Added Value of Systemic Lidocaine on Postoperative Pain, Opiate Use and Nausea After Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMS.2017.032
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Surgery; Pain, Postoperative; Nausea, Postoperative; Opioid Use
Keywords: postoperative analgesia; knee surgery; intravenous lidocaine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Group A receives linisol 2%, group B receives placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medicine used for each individual patient will be prepared by the nurse not otherwise involved in patient data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic lidocaine (Active Comparator): Lidocaine 2% IV bolus: 1.5 mg/kg at induction of anesthesia and at the end of surgery.
  Interventions: Drug: systemic lidocaine
- Placebo (Placebo Comparator): Saline 0.9% IV bolus: 0.075 ml/kg at induction of anesthesia and at the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: systemic lidocaine — Systemic lidocaine is administrated at induction of anesthesia and at the end of surgery (1.5 mg/kg).
  Other Names: linisol 2%
  Arms: systemic lidocaine
Drug: Placebo — Placebo is administrated at induction of anesthesia and at the end of surgery (0.075 ml/kg)
  Other Names: saline 0.9%
  Arms: Placebo

SUMMARY:
Local intra-articular injection of anesthetics (LIA) is increasingly used during knee arthroscopy for pain relief. The LIA can only be performed at the end of surgery as the knee joint is continuously flushed during the arthroscopy. As a consequence, an optimal analgesic effect is only obtained one hour after surgery and opiates are typically used as pain relief in the immediate postoperative period. Since these opiates have a number of side effects such as nausea, vomiting and drowsiness, other analgetic methods are desirable.

Intravenous administration of lidocaine, a safe, inexpensive analgesic, is already used in major (abdominal) surgeries and might also be a promising method for pain relief in the first hour after knee arthroscopy, in anticipation of the onset of the analgesic effect of the LIA.

The aim of this study is to verify if systemic administration of lidocaine has a beneficial effect on the pain immediately after knee arthroscopy. In addition, the effect of systemic lidocaine administration on postoperative nausea, vomiting and general patient comfort will be evaluated.

DETAILED DESCRIPTION:
2X30 patients which are planned for elective knee arthroscopy are randomised: Lidocaine-group and Placebo-group.

All patients receive standardised multimodal intravenous analgesia. After standardised induction of anesthesia, patient positioning and administration of basic analgetics paracetamol & diclofenac, the patient is administered either linisol 2% (1.5 mg/kg) or placebo NaCl 0.9% (0.075 ml/kg = equivalent volume). At the end of the procedure, linisol or placebo is readministered at the same dose. The surgeon and anesthesiologist are blinded for patient allocation.

Postoperative analgesic consumption, nausea and vomiting (PONV), general comfort and pain scores are recorded. Visual Analogue scores (VAS) for knee pain are assessed before surgery, 1-15 minutes after awakening, at the moment of discharge from the post-anesthesia care unit (PACU) and at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients which are planned for elective knee arthroscopy
* ASA 1 and 2
* knee arthroscopy suitable for intra-articular injection of anesthetics

Exclusion Criteria:

* contra-indication for lidocaine, paracetamol or diclofenac
* known history of severe post-operative nausea or vomiting
* knee arthroscopy associated with anterior cruciate ligament reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score for pain | from moment of surgery until hospital discharge. on average 8 hours after surgery
  Pain intensity using the VAS, where 0 = no pain and 100 = pain as bad as can be) before surgery, 1-15 minutes after awakening, at discharge from the PACU and from the hospital

SECONDARY OUTCOMES:
incidence of Nausea and vomiting | from moment of surgery until hospital discharge. on average 8 hours after surgery
  Incidence of postoperative nausea and vomiting
PONV treatment | from moment of surgery until hospital discharge. on average 8 hours after surgery
  Number of pharmacological treatments for Postoperative Nausea & Vomiting (PONV)
opioid use | at the PACU on average 60 minutes
  dosing and frequency of opioid use
length of stay at the PACU | from moment of surgery until discharge from the PACU. on average 60 minutes after surgery
  Time (in minutes) between the end of surgery and the discharge from the PACU
general patient comfort | at the moment before of hospital discharge. on average 8 hours after surgery.
  VAS for general comfort : from 0 until 100 (0= extremely dissatisfied ; 100= extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD,PhD,MSc, Principal Investigator — Maria Middelares Hospital
Locations (1):
- AZ Maria Middelares, Ghent, Oost, Belgium

IPD SHARING:
Plan to Share IPD: Undecided